CLINICAL TRIAL: NCT05333081
Title: Determination of the Glycemic Index of 25 Italian Rice Varieties
Brief Title: Glycemic Index of Italian Rice Varieties
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0107/11012022
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Glycemic Index

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of the glycemic index (Other)
  Interventions: Other: Consumption of rice for evaluation of the glycemic index

INTERVENTIONS:
Other: Consumption of rice for evaluation of the glycemic index — The test of each food was carried out for a maximum time of 120 minutes, by carrying out repeated measurements of the glycaemia of all subjects at a distance of 0, 15, 30, 45, 60, 90 and 120 minutes from the administration of the sample in order to obtain a glycemic curve for each sample considered.

SUMMARY:
The service commissioned by the National Rice Authority required the evaluation of the Glycemic Index of 25 varieties of rice. As a reference, both for the comparison and for the calculation of the Glycemic Index, glucose was used, which clearly has characteristics of greater uniformity than white bread and was preferred because it is better suited to be used as a standard of measurement. In accordance with the ISO 26642 standard, a panel of selected volunteers (consisting of 10 subjects), healthy, not suffering from diabetes or other pathologies of glucose metabolism, were included in the study. As per protocol, the changes in glycaemia of all the subjects involved were evaluated after the intake of glucose (50g), as a standard food, and of rice (50g of available carbohydrates), taking into account the carbohydrate content of each variety. to determine the amount of rice to be fed. The test of each food was carried out for a maximum time of 120 minutes, by carrying out repeated measurements of the glycaemia of all subjects at a distance of 0, 15, 30, 45, 60, 90 and 120 minutes from the administration of the sample in order to obtain a glycemic curve for each sample considered.

From the analysis of the area underlying the glycemic curve of each variety, it was possible to determine the Glycemic Index.

ELIGIBILITY:
Inclusion Criteria:

* no known foood allergy or intolerance
* no medications to affect glucose tolerance

Exclusion Criteria:

* Diabetes mellitus or insulin disorders
* major event or surgical procedure requiring hospitalization within the preceding 3 months
* disease or drugs that influcence digestion and absorbtion of nutrients
* the use of steroids, protease inhibitors or antipsychotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of glucose response | From baseline to 120 min after rice consumption
  Gycemia (mg/dl)

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda di Servizi alla Persona, Pavia, Italy

REFERENCES:
- [Derived] Rondanelli M, Ferrario RA, Barrile GC, Guido D, Gasparri C, Ferraris C, Cavioni A, Mansueto F, Mazzola G, Patelli Z, Peroni G, Pirola M, Razza C, Tartara A, Perna S. The Glycemic Index of Indica and Japonica Subspecies Parboiled Rice Grown in Italy and the Effect on Glycemic Index of Different Parboiling Processes. J Med Food. 2023 Jun;26(6):422-427. doi: 10.1089/jmf.2022.0120. Epub 2023 Jun 1. PMID 37262189